CLINICAL TRIAL: NCT02566824
Title: A Cognitive Behavioral Therapy Group Intervention for Adolescents With Attention-Deficit / Hyperactivity Disorder
Brief Title: Cognitive Behavioral Therapy for Adolescents With Attention-Deficit / Hyperactivity Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lily Hechtman, Professor of Psychiatry and Pediatrics; Director of Research - Division of Child Psychiatry, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED-05-055
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics; Methylphenidate; Dextroamphetamine; SLI381; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavioural & Skills Training (Experimental): Participants can choose to be on medication or not. If they decide to take medication, they will be titrated to an optimal dose of stimulant medication. Then they undergo the 12 weeks of group cognitive behavioral and skills training therapy.
  Interventions: Behavioral: Cognitive Behavioural & Skills Training; Drug: Methylphenidate or amphetamine product
- Supportive Group Therapy (Active Comparator): Participants can choose to be on medication or not. If they decide to take medication, they will be titrated to an optimal dose of stimulant medication. Then they undergo the 12 weeks of supportive group therapy.
  Interventions: Behavioral: Supportive Group Therapy; Drug: Methylphenidate or amphetamine product
- Treatment as Usual - community resources (Active Comparator): Participants can choose to be on medication or not. If they decide to take medication, they will be titrated to an optimal dose of stimulant medication. Then they are referred to their treating physicians and are free to use any resources that are available to them in their communities.
  Interventions: Other: Treatment as Usual - community resources; Drug: Methylphenidate or amphetamine product

INTERVENTIONS:
Behavioral: Cognitive Behavioural & Skills Training — This will be administered in groups of 10 participants in 12 sessions each lasting 1.5 hours. Each session will focus on a new topic- Modules will be introduced via role play illustrating the topic, followed by Q&A. Strategies will be introduced to address the problems illustrated. Adolescents will practice using these strategies via planned activities or games. Obstacles to applying the skills in everyday life will be discussed and a physical reminder will be provided for each skill. A homework activity will be assigned to help participants practice the skill during the week. Each session will begin with homework review. Adolescents will also receive individual telephone coaching twice a week during the 12 weeks, which will taper off during the follow-up phase. Parents will also attend their own support group.
  Arms: Cognitive Behavioural & Skills Training
Behavioral: Supportive Group Therapy — This will be administered in groups of 10 participants in 12 sessions each session lasting 1.5 hours. During the initial session group members will be asked to identify a specific goal to address during the program. Each session will review the previous week's events (challenges and positive accomplishments) and psychoeducation on a topic relating to ADHD (topics will be elicited from group members at the outset of each session). Adolescents will also receive a telephone coaching at the same frequency as the CBT+S group participants. These phone calls will deal with issues a given participant had raised in the preceding session, and the approach will emphasize support and unconditional positive regard. Parents will also attend their own support group.
  Arms: Supportive Group Therapy
Other: Treatment as Usual - community resources — The treatment as usual group reflects what patients currently receive in the community (mainly medication). Participants will be stabilized on optimal medication (if they choose to be on medication) and referred back to the community for follow-up. Participants are free to seek out any additional interventions that they feel are required. These participants will be evaluated at the same intervals as the two therapy groups. They will receive a follow-up phone call from the study coordinator at two-month intervals in-between evaluation points. If participants indicate during the phone call that they require services, they will be referred to services in the community.
  Arms: Treatment as Usual - community resources
Drug: Methylphenidate or amphetamine product — Medication is titrated over a 4-week period with stepwise increments each week. Participants, parents and teachers complete ADHD symptom scales at baseline and before each medication visit. They will also complete side effects scales at baseline and before each medication visit. The gradual increase will continue until there is no further improvement in symptoms and in the Clinical Global Improvement Scale or side effects are such that further increases are not indicated. Once the optimal dose is reached, the participants remain on this dose for the remainder of the study.
  Other Names: Ritalin; Concerta; Biphentin; Dexedrine; Adderall XR; Vyvanse

SUMMARY:
Attention Deficit/ Hyperactivity Disorder (ADHD) is a common childhood psychiatric condition, which often persists into adolescence. In adolescence ADHD is associated with poor academic, social, and emotional functioning, other psychiatric problems, substance abuse, and antisocial behaviour. Although medication effectively reduces symptoms such as hyperactivity and inattention, it does not directly address academic, social, emotional, and behavioural problems. Overcoming these would require building skills in organization, time management, problem solving, emotional modulation, stress management and interpersonal rapport. Yet, psychosocial treatments targeting such skills in adolescents with ADHD have been little studied and are scarce in the community. The proposed study will evaluate cognitive behavioural and skills training therapy (CBT+S) for adolescents with ADHD. Adolescents will decide whether they want to take medication to treat their ADHD symptoms. If they choose to be on medication, they will be stabilized on optimized medication and randomly assigned to 12 sessions of either manualized group cognitive behavioral and skills training therapy (CBT+S) or manualized supportive group therapy (SGT). An additional treatment-as-usual group will also be included. CBT+S will focus on skill acquisition in common problem areas for adolescents with ADHD, such as organization and time management, distractibility, impulsivity, and social skills. A coach will call each participant twice a week to help practice the learned skills.

Parallel groups will be provided for parents of CBT+S and SGT participants focusing on education, support and sharing experiences. If CBT+S proves to benefit adolescents with ADHD, it can be made widely available to these adolescents in the community. This would help them improve their academic, social, and emotional functioning and ultimately their long term outcomes.

DETAILED DESCRIPTION:
Attention Deficit/ Hyperactivity Disorder (ADHD) is a prevalent childhood psychiatric condition affecting 5-10% of children worldwide. ADHD persists into adolescence in 70-80% of those diagnosed in childhood. In adolescence, ADHD is associated with impairments in academic, social, and emotional functioning, as well as with elevated rates of psychiatric comorbidities, substance abuse, and antisocial behaviour.

Medication is currently the mainstay treatment for adolescents with ADHD. Although medication is an efficacious treatment for core ADHD symptoms, it does not directly address the associated academic, social, emotional and behavioural impairments. Overcoming these would require skills in organization, time management, problem solving, emotional modulation, stress management and interpersonal rapport. While these skills are important in childhood, they become particularly indispensable as the child enters adolescence and is expected to function more autonomously. However, little is known about the efficacy of psychosocial treatments targeting such skills for adolescents with ADHD, and there are few psychosocial treatment options available to these adolescents in the community.

The purpose of the study will be to evaluate the efficacy of a novel integrative therapy that uses cognitive-behavioural approaches to foster the development of these skills in adolescents with ADHD. Adolescents with ADHD, ages 13-17, will be randomly assigned to either 12 sessions of manualized group cognitive behavioural and skills training therapy (CBT+S) or to 12 sessions of manualized supportive group therapy (SGT). The CBT+S sessions will focus on acquisition of skills targeting the common functional deficits of adolescents with ADHD, with the modules covering psychoeducation, goal attainment, organization, time management, focus training and distractibility reduction, impulse control, study skills, stress management, cognitive restructuring, anger management, social skills, and self-esteem. A coach will call each participant twice a week to help implement CBT+S strategies in daily life. Supportive group therapy (SGT) for the adolescents will focus on increasing understanding of ADHD, sharing experiences, and fostering a network of support. Calls from a coach will deal with participant-elicited issues. Parents of all adolescents will participate in parallel 6-session support groups similar to SGT and focused on psychoeducation, sharing and support. Treatment effects will be evaluated after 12 weeks of treatment. Maintenance of treatment benefits will be evaluated after 4 and 8 months of follow up. A treatment as usual group will be used to control for repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 17 years
* The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) ADHD diagnosis confirmed by a psychiatrist
* Intelligent Quotient (IQ) > 80 as per the Wechsler Intelligence Scale for Children -Fifth Edition (WISC-V)

Exclusion Criteria:

* History of Pervasive Development Disorder (PDD) or psychosis
* Significant brain traumas (encephalitis, head injury, etc.)
* Major medical conditions or impairments that would interfere with the ability of the adolescent to complete testing or take psychostimulants, e.g., epilepsy, cardiac abnormalities, or renal abnormalities
* Significant psychiatric comorbidities (e.g. suicidality) or substance abuse requiring immediate treatment.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2010-10; Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit/Hyperactivity Disorder (ADHD) Symptomatology (measured via Conners' 3 Adolescent Self-Report Scale short form; Conners' 3 parent version; Conners' 3 teacher version) - Change from baseline | At baseline - once medication is optimally titrated (if medication is chosen)
Attention Deficit/Hyperactivity Disorder (ADHD) Symptomatology (measured via Conners' 3 Adolescent Self-Report Scale short form; Conners' 3 parent version; Conners' 3 teacher version) - Change from baseline | After 12 weeks of group treatment or 12 weeks after medication has been optimally titrated (if medication is chosen)
Attention Deficit/Hyperactivity Disorder (ADHD) Symptomatology (measured via Conners' 3 Adolescent Self-Report Scale short form; Conners' 3 parent version; Conners' 3 teacher version) - Change from baseline | Four months after the end of group treatment or 7 1/2 months after medication has been optimally titrated (if medication is chosen)
Attention Deficit/Hyperactivity Disorder (ADHD) Symptomatology (measured via Conners' 3 Adolescent Self-Report Scale short form; Conners' 3 parent version; Conners' 3 teacher version) - Change from baseline | Eight months after the end of group treatment or 11 1/2 months after medication has been optimally titrated (if medication is chosen)

SECONDARY OUTCOMES:
Organizational skills (measured via Children's Organizational Skills Scale (COSS) completed by adolescent and parent) - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Emotional adjustment - (including ODD, conduct disorder symptoms, depression, and anxiety) measured via Stony Brook Child and Adolescent Symptom Inventory - 5 (CASI-5) completed by adolescent and parent - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Self-esteem - evaluated via Rosenberg Self Esteem Scale (RSES) completed by the adolescent - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Social skills measured via Social Skills Improvement System (SSIS) completed by adolescent and parent - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Parent-adolescent conflict measured via the Parent Issues Checklist- Revised completed by the parent - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated

OTHER OUTCOMES:
Global functional impairment measured using Weiss Functional Impairment Rating Scale (WFIRS) completed by the adolescent and the parent - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Global functional impairment measured via Sheehan Disability Scale, completed by adolescent, parent, and a blind clinician - Change from baseline | At baseline - optimally titrated(if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated
Global functional impairment measured via Clinical Global Impression Scale (CGI) completed by a blind clinician - Change from baseline | At baseline - optimally titrated (if medicated); after group treatment or 12 weeks after optimally titrated; 4 months after group treatment or 7 1/2 months after optimally titrated; 8 months after group treatment or 11 1/2 months after optimally titrated

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hechtman, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available.